CLINICAL TRIAL: NCT02548949
Title: KOREAN POST MARKETING SURVEILLANCE TO OBSERVE EFFECTIVENESS AND SAFETY OF PRISTIQ (REGISTERED) IN PATIENTS WITH MAJOR DEPRESSIVE DISORDER.
Brief Title: Korean Post Marketing Surveillance to Observe Effectiveness and Safety of PRISTIQ
Acronym: PMS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B2061143
Record Dates: First submitted 2015-07-16; First posted 2015-09-14 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — Retention of biospecimen is not needed necessarily. If the investigator check blood sample under routine practice during the study, investigator record results of blood sampling, such as CBC and blood chemistry.
  Full lists of recordings are following : Hemoglobin, Hematocrit, RBC, WBC, Platelets, Sodium, Potassium, BUN, Creatinine, Calcium, Total Bilirubin, SGOT/AST, SGPT/ALT, Cholesterol.
Oversight: Data Monitoring Committee: No

SUMMARY:
On 6 Feb 2014, Pristiq was approved for the treatment of Major Depressive Disorder(MDD) in Korea. In accordance with the Standards for Re-examination of New Drug, it is required to conduct a PMS for 600 patients by 5 Feb 2020. Post marketing surveillance is required to determine any problems or questions associated with Pristiq after marketing, with regard to the following clauses under conditions of general clinical practice. Therefore, through this study, effectiveness and safety of pristiq will be observed.

DETAILED DESCRIPTION:
The objective of this study is to determine any problems or questions associated with Pristiq after marketing, with regard to the following clauses under conditions of general clinical practice, in compliance with the regulation "Re-examination guideline of new drugs (Ministry of Food and Drug Safety Notification 2013-251, 2013.12.20)".

1. Serious adverse event/adverse drug reaction
2. Unexpected adverse event/adverse drug reaction that have not been reflected in the approved drug label.
3. Known adverse drug reaction
4. Non-serious adverse drug reaction
5. Other safety and effectiveness information

ELIGIBILITY:
Inclusion Criteria:

1. Adults 19 years of age or older, who have been received at least one dose of PRISTIQ® for the treatment of Major depressive disorder (MDD).
2. Patients who have been received for the first time after signed the 'data privacy statement'

Exclusion Criteria:

Patients to whom PRISTIQ® is contraindicated as per the local labeling;

1. Hypersensitivity to desvenlafaxine succinate, venlafaxine hydrochloride or any excipients in the PRISTIQ® formulation.
2. Serotonin syndrome and MAOIs: Do not use MAOIs intended to treat psychiatric disorders with PRISTIQ® or Do not use PRISTIQ® within 14 days of stopping an MAOI intended to treat psychiatric disorders

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 19 years of age or older, who have been received at least one dose of PRISTIQ® for the treatment of Major depressive disorder (MDD). The study population would be enrolled in multi-center in which subjects are administered PRISTIQ as part of routine practice at Korean health care centers by accredited psychiatrists.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- South Korea (22):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheonbuk-do
  - Hallym University Dongtan Sacred Heart Hospital/Department of Neuropsychiatry, Hwaseong-si, Gyeonggi Province
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Roa Neurology Clinic/Neurology, Bundang-gu, Seongnam-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Bundang Cha Medical Center, Seongnam-si, Gyeonggi-do
  - Konkuk University Chungju Hospital / Department of Psychiatry, Chungju, North Chungcheong
  - Bong Seng Memorial Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chuncheon Sacred Heart Hospital-Hallym University, Gangwon-do
  - Chosun University Hospital, Gwangju
  - Chonnam National University Hospital, Gwangju
  - Presbyterian Medical Center, Jeonju
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong Department of Psychiatry, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Roh S, Lee KS, Choi S, Kim JM. Safety and Effectiveness of Desvenlafaxine in Korean Patients with Major Depressive Disorder: A 6-month Postmarketing Surveillance Study. Clin Psychopharmacol Neurosci. 2022 Aug 31;20(3):548-559. doi: 10.9758/cpn.2022.20.3.548. PMID 35879039
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B2061143

RESULTS

PARTICIPANT FLOW:
Groups:
- Pristiq: Participants who were receiving Pristiq tablets as part of routine practice at Korean health care centers were enrolled and observed in this study for up to 8 weeks since the start of Pristiq administration.
Period: Overall Study
Arm/Group | Pristiq
Started | 700
Completed | 700
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had been administered Pristiq at least once and completed follow up.
Arm/Group | Pristiq
Number analyzed (Participants) | 700
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.23 (17.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455
  Male | 245
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 8 weeks
Population: Safety analysis set included all participants who had been administered Pristiq at least once and completed follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristiq
Number analyzed (Participants) | 700
Participants
  AEs | 80
  SAEs | 3

2. Primary Outcome: Number of Participants in Each Category of Clinical Global Impression-Improvement (CGI-I) Scale
Description: CGI-I scale was a 7-point scale used to assess clinical effectiveness on a range of 1 to 7; where, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = No change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Higher score indicated worse condition/lower clinical effectiveness.
Time Frame: At Week 8
Population: Effectiveness analysis set included all participants who had been administered Pristiq at least once and were evaluated upon its related effectiveness outcomes at least once. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristiq
Number analyzed (Participants) | 454
Participants
  Very much improved | 22
  Much improved | 128
  Minimally improved | 237
  No change | 65
  Minimally worse | 2
  Much worse | 0
  Very much worse | 0

3. Primary Outcome: Number of Participants With Final Effectiveness Evaluation
Description: Final effectiveness was evaluated as 'improved', 'no change', 'worse' or 'unevaluable' based on overall participant's clinical response after 8 weeks of Pristiq administration (as part of routine care), where, Improved = there was the improvement of symptoms related to major depressive disorder, No change = there was no significant change compared to participant's status before Pristiq administration, Worse = symptoms were getting worse compared to participant's status before Pristiq administration, Unevaluable = the medical charts do not had adequate progress notes to make a judgment on clinical response.
Time Frame: At Week 8
Population: Effectiveness analysis set included all participants who had been administered Pristiq at least once and were evaluated upon its related effectiveness outcomes at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristiq
Number analyzed (Participants) | 479
Participants
  Improved | 411
  No change | 68
  Worse | 0
  Unevaluable | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety analysis set included all participants who had been administered Pristiq at least once and completed follow up.
Arm/Group | Pristiq
All-Cause Mortality (participants affected / at risk) | 0/700
Serious Adverse Events (participants affected / at risk) | 3/700
Other Adverse Events (participants affected / at risk) | 80/700
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pristiq (N=700)
Chest pain (General disorders) | 1
Angina pectoris aggravated (Cardiac disorders) | 1
Tremor (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pristiq (N=700)
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Fever (General disorders) | 2
Medicine ineffective (General disorders) | 1
Oedema generalised (General disorders) | 1
Hypertension (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 4
Arthritis rheumatoid aggravated (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Appetite decreased (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
Enteritis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastroesophageal reflux (Gastrointestinal disorders) | 1
Mouth dry (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 14
Oesophagitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Palpitation (Cardiac disorders) | 4
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 4
Globus hystericus (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 6
Somnolence (Psychiatric disorders) | 10
Thinking abnormal (Psychiatric disorders) | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Diaphoresis (Skin and subcutaneous tissue disorders) | 2
Dysuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT02548949/SAP_000.pdf
  • Study Protocol (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT02548949/Prot_001.pdf